CLINICAL TRIAL: NCT00031148
Title: Phase I/II Trial of Keratinocyte Growth Factor (rHuKGF) to Prevent Acute GVHD in 6/6 HLA=BMT Recipients
Brief Title: Keratinocyte Growth Factor to Prevent Acute GVHD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: FD-R-2021-01; FD-R-002021-01
Record Dates: First submitted 2002-02-26; First posted 2002-02-27 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2002-01

CONDITIONS: Graft-vs-Host Disease
Keywords: Keratinocyte growth factor; Bone Marrow Transplantation; Hematopoietic Stem Cell Transplantation; HLA Antigens; Transplantation, Homologous; Recombinant Proteins
MeSH Terms: conditions — Graft vs Host Disease | interventions — Fibroblast Growth Factor 7

INTERVENTIONS:
Drug: Recombinant Human Keratinocyte Growth Factor (rHuKGF)

SUMMARY:
This is a study to determine the safety and efficacy of keratinocyte growth factor (KGF) to prevent acute graft-versus-host disease (GVHD) in patients undergoing allogeneic bone marrow (BM) or peripheral blood progenitor cell (PBPC) transplantation.

DETAILED DESCRIPTION:
GVHD remains the major complication of allogeneic BM transplantation and is initiated during the conditioning of the recipient for transplant when the host tissues are damaged. Research has demonstrated that the gastrointestinal (GI) tract is a critical organ in GVHD pathophysiology. Agents that protect the GI tract may provide prophylaxis against the cytokine cascade and can lead to a reduced incidence and severity of GVHD. KGF is a protein that stimulates the growth of epithelial cells including those of the GI tract. KGF can protect the GI tract, prevent GVHD, and preserve donor T-cell function.

Patients will receive standard GVHD prophylaxis in addition to the study drug. Overall GVHD will be graded weekly during the first 2 months after transplant, then every other week to Day 100. Response to therapy will be measured through the use of severity indices, physical exam, and laboratory serum values.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of a hematological malignancy, including myelodysplastic syndromes.
* Eligible for cyclophosphamide and total body irradiation conditioning therapy or busulphan and cyclophosphamide conditioning therapy.
* Must have a 6/6 human leukocyte antigens (HLA)-matched family member donor.
* Women must be post-menopausal, sterile, or using effective contraception for 1 month before, during, and for 2 months after study.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.

Exclusion criteria:

* T-cell depletion for GVHD prophylaxis.
* Active hepatitis.
* Pre-existent inflammatory bowel disease requiring active therapy.
* Active uncontrolled infection.
* Prior bone marrow or peripheral blood stem cell (PBSC) transplantation.
* Documented hypersensitivity to rHuKGF.
* Prior enrollment to a study of rHuKGF.
* HIV-positive.
* Pregnant or nursing.
* Active chronic skin disease requiring therapy.

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72
Dates: Start 2001-09; Study Completion 2003-08

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan Cancer Center, Ann Arbor, Michigan, United States